CLINICAL TRIAL: NCT01130168
Title: A Double-Blind, Randomized, Placebo-Controlled, 3-Period, Crossover Study to Evaluate the Effects of Antihypertensive Agents on Central Blood Pressure in Healthy Subjects and Patients With Hypertension
Brief Title: The Effects of Antihypertensive Agents on Central Blood Pressure in Healthy Participants and Participants With Hypertension (MK-0000-166) (COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-166; 2010_537
Record Dates: First submitted 2010-05-19; First posted 2010-05-25 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo/ISMN ER/Amlodipine (Sequence 1) (Experimental): Participants received a dose-matched Placebo capsule orally for 4 weeks during Period 1, followed by a ISMN ER 30 mg capsule orally for 4 weeks during Period 2, followed by Amlodipine 10 mg (two 5 mg capsules) orally for 4 weeks during Period 3, with a 2-week washout between each period.
  Interventions: Drug: Placebo; Drug: Comparator: Amlodipine; Drug: Comparator: ISMN ER
- ISMN ER/Amlodipine/Placebo (Sequence 2) (Experimental): Participants received a ISMN ER 30 mg capsule orally for 4 weeks during Period 1, followed by Amlodipine 10 mg (two 5 mg capsules) orally for 4 weeks during Period 2, followed by a dose-matched Placebo capsule orally for 4 weeks during Period 3, with a 2-week washout between each period.
  Interventions: Drug: Placebo; Drug: Comparator: Amlodipine; Drug: Comparator: ISMN ER
- Amlodipine/Placebo/ISMN ER (Sequence 3) (Experimental): Participants received Amlodipine 10 mg (two 5 mg capsules) orally for 4 weeks during Period 1, followed by a dose-matched Placebo capsule orally for 4 weeks during Period 2, followed by a ISMN ER 30 mg capsule orally for 4 weeks during Period 3, with a 2-week washout between each period.
  Interventions: Drug: Placebo; Drug: Comparator: Amlodipine; Drug: Comparator: ISMN ER
- ISMN ER/Placebo/Amlodipine (Sequence 4) (Experimental): Participants received a ISMN ER 30 mg capsule orally for 4 weeks during Period 1, followed by a dose-matched Placebo capsule orally for 4 weeks during Period 2, followed by Amlodipine 10 mg (two 5 mg capsules) orally for 4 weeks during Period 3, with a 2-week washout between each period.
  Interventions: Drug: Placebo; Drug: Comparator: Amlodipine; Drug: Comparator: ISMN ER
- Placebo/Amlodipine/ISMN ER (Sequence 5) (Experimental): Participants received a dose-matched Placebo capsule orally for 4 weeks during Period 1, followed by Amlodipine 10 mg (two 5 mg capsules) orally for 4 weeks during Period 2, followed by a ISMN ER 30 mg capsule orally for 4 weeks during Period 3, with a 2-week washout between each period.
  Interventions: Drug: Placebo; Drug: Comparator: Amlodipine; Drug: Comparator: ISMN ER
- Amlodipine/ISMN ER/Placebo (Sequence 6) (Experimental): Participants received Amlodipine 10 mg (two 5 mg capsules) orally for 4 weeks during Period 1, followed by a ISMN ER 30 mg capsule orally for 4 weeks during Period 2, followed by a dose-matched Placebo capsule for 4 weeks during Period, with a 2-week washout between each period.
  Interventions: Drug: Placebo; Drug: Comparator: Amlodipine; Drug: Comparator: ISMN ER

INTERVENTIONS:
Drug: Placebo — Placebo, capsule taken orally once daily during 4 weeks of treatment
Drug: Comparator: Amlodipine — Amlodipine 10 mg, taken orally as two 5 mg capsules, single daily dose for 4 weeks
Drug: Comparator: ISMN ER — ISMN ER 30 mg capsule, taken orally as single daily dose for 4 weeks

SUMMARY:
This study will test the relationship between CBP (central blood pressure) and PBP (peripheral blood pressure) effects after single and multiple doses of Isosorbide mononitrate extended release (ISMN ER) or Amlodipine besylate in participants with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a male or female between 30 and 65 years of age (inclusive) at the pre-study (screening)
* Female participant of childbearing potential must have a negative pregnancy test
* Participant has a brachial systolic blood pressure >130 mm Hg

and <180 mm Hg

* Participant has a Body Mass Index (BMI) that is >20 kg/m^2 and <35 kg/m^2
* Participant has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months

Exclusion Criteria:

* Female Participant is pregnant or lactating
* Participant anticipates the use of Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) other than acetaminophen
* Participant is currently a user (including "recreational use") of any illicit drugs, has a history of drug or alcohol abuse within approximately 2 years, or has a positive prestudy urine drug screen
* Participant has a condition for which there is a warning, contraindication, or precaution against the use of ISMN ER including: acute myocardial infarction or congestive heart failure, hypotension, volume depletion, and pregnancy
* Participant has a history of significant drug allergy or any clinically significant adverse experience of a serious nature related to the administration of either a marketed or an investigational drug, including nitrates, nitrites, Amlodipine, and ISMN ER

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/ISMN ER/Amlodipine (Sequence 1): Participants received a dose-matched Placebo capsule orally for 4 weeks during Period 1, followed by a ISMN ER 30 mg capsule orally for 4 weeks during Period 2, followed by Amlodipine 10 mg (two 5 mg capsules) orally for 4 weeks during Period 3, with a 2-week washout between each period. Experimental: ISMN ER/Amlodipine/Placebo
Period: Period 1
Arm/Group | Placebo/ISMN ER/Amlodipine (Sequence 1) | ISMN ER/Amlodipine/Placebo (Sequence 2) | Amlodipine/Placebo/ISMN ER (Sequence 3) | ISMN ER/Placebo/Amlodipine (Sequence 4) | Placebo/Amlodipine/ISMN ER (Sequence 5) | Amlodipine/ISMN ER/Placebo (Sequence 6)
Started | 6 | 7 | 6 | 8 | 5 | 6
Completed | 6 | 6 | 5 | 5 | 5 | 6
Not Completed | 0 | 1 | 1 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Discontinued For Other Reason | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 2
Arm/Group | Placebo/ISMN ER/Amlodipine (Sequence 1) | ISMN ER/Amlodipine/Placebo (Sequence 2) | Amlodipine/Placebo/ISMN ER (Sequence 3) | ISMN ER/Placebo/Amlodipine (Sequence 4) | Placebo/Amlodipine/ISMN ER (Sequence 5) | Amlodipine/ISMN ER/Placebo (Sequence 6)
Started | 6 | 6 | 5 | 5 | 5 | 6
Completed | 6 | 6 | 5 | 5 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Placebo/ISMN ER/Amlodipine (Sequence 1) | ISMN ER/Amlodipine/Placebo (Sequence 2) | Amlodipine/Placebo/ISMN ER (Sequence 3) | ISMN ER/Placebo/Amlodipine (Sequence 4) | Placebo/Amlodipine/ISMN ER (Sequence 5) | Amlodipine/ISMN ER/Placebo (Sequence 6)
Started | 6 | 6 | 5 | 5 | 5 | 6
Completed | 6 | 6 | 5 | 5 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] — Age data were not reported for 5 participants who were excluded from analysis.
  years | 49 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender data were not reported for 5 participants who were excluded from analysis.
  Participants
    Female | 11
    Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Average (TWA) Change From Baseline (0 Hours) to 12 Hours in Heart-Rate-Corrected Augmentation Index (AIx) After A Single Dose of Treatment
Description: The augmentation index (AIx) is a measure of systemic arterial stiffness, and is the ratio of augmented aortic pressure (Δ P) to central pulse pressure expressed as a percent. AIx = (ΔP/PP) x 100, where P = pressure and PP = Pulse Pressure. Single dose effects on AIx were estimated as a time-weighted average change from baseline over the 12-hour post single dose observation period. Because heart rate (HR) affects AIx, AIx was corrected to a HR of 75 beats per minute (bpm) as follows:
  HR-corrected AIx = -0.39 x (75 - HR) + AIx. This value was used for all AIx analyses.
Time Frame: Baseline (0 hrs), 12 hours post-dose (Day 1)
Population: 33 participants completed all study periods and provided more than 1 period of BP data, and were thus evaluable for the BP analyses.
  Unreliable SphygmoCor® data were collected for one participant in the ISM ER treatment group, therefore this participant was excluded from the single dose AIx analysis.
Measure: Least Squares Mean (Standard Deviation); unit: percent
Groups:
- ISMN ER: Isosorbide mononitrate extended release (ISMN ER) was administered as a 30 mg single daily dose over 4 weeks.
- Amlodipine: Amlodipine was administered as a 10 mg single daily dose over 4 weeks.
- Placebo: Placebo was administered as a single once daily dose during 4 weeks of treatment.
Arm/Group | ISMN ER | Amlodipine | Placebo
Number analyzed (Participants) | 32 | 33 | 33
percent | -11.1 (4.5) [-22.0 to 4.0] | -0.7 (4.5) [-13.0 to 8.0] | 2.1 (4.5) [-6.0 to 10.0]
Statistical Analysis 1: Comparison: ISMN ER vs Placebo; Test type: Superiority or Other; p < 0.0005, ANOVA; Mean Difference (Final Values) = -13.1, 95% CI 2-sided [-15.3 to -10.9]
Statistical Analysis 2: Comparison: Amlodipine vs Placebo; Test type: Superiority or Other; p = 0.016, ANOVA; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-4.9 to -0.6]

2. Primary Outcome: Change From Baseline (0 Hours) to Week 4 in Heart-Rate-Corrected AIx After Multiple Doses of Treatment
Description: The augmentation index (AIx) is a measure of systemic arterial stiffness, and is the ratio of augmented aortic pressure (Δ P) to central pulse pressure expressed as a percent. AIx = (ΔP/PP) x 100, where P = pressure and PP = Pulse Pressure. Because heart rate (HR) affects AIx, AIx was corrected to a HR of 75 beats per minute (bpm) as follows:
  HR-corrected AIx = -0.39 x (75 - HR) + AIx. This value was used for all AIx analyses.
Time Frame: Baseline (0 hrs), 24 hours after the Day 28 dose
Population: 33 participants completed all study periods and provided more than 1 period of BP data, and were thus evaluable for the BP analyses.
  Unreliable SphygmoCor® data were collected for two participants in the ISM ER treatment group, therefore these participants were excluded from the multiple dose AIx analysis.
Measure: Least Squares Mean (Standard Deviation); unit: percent
Groups:
- ISMN ER: ISMN ER was administered as a 30 mg single daily dose over 4 weeks.
Arm/Group | ISMN ER | Amlodipine | Placebo
Number analyzed (Participants) | 31 | 33 | 33
percent | 2.5 (6.2) | -4.7 (6.2) | 1.2 (6.2)
Statistical Analysis 1: Comparison: ISMN ER vs Placebo; Test type: Superiority or Other; p = 0.407, ANOVA; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-1.7 to 4.3]
Statistical Analysis 2: Comparison: Amlodipine vs Placebo; Test type: Superiority or Other; p < 0.0005, ANOVA; Mean Difference (Final Values) = -5.9, 95% CI 2-sided [-8.9 to -2.9]

3. Primary Outcome: TWA Change From Baseline (0 Hours) to 12 Hours in Central Systolic Blood Pressure (SBP) After A Single Dose of Treatment
Description: Central SBP was measured by the SphygmoCor® device. Single dose effects on central SBP were estimated as a time-weighted average change from baseline over the 12-hour post single dose observation period.
Time Frame: Baseline (0 hrs), 12 hours post-dose (Day 1)
Population: 33 participants completed all study periods and provided more than 1 period of BP data, and were thus evaluable for the BP analyses.
  Unreliable SphygmoCor® data were collected for one participant in the ISM ER treatment group, therefore this participant was excluded from the single dose SBP analysis.
Measure: Least Squares Mean (Standard Deviation); unit: mm mercury (Hg)
Arm/Group | ISMN ER | Amlodipine | Placebo
Number analyzed (Participants) | 32 | 33 | 33
mm mercury (Hg) | -14.7 (7.7) | -3.6 (7.7) | 2.7 (7.7)
Statistical Analysis 1: Comparison: ISMN ER vs Placebo; Test type: Superiority or Other; p < 0.0005, ANOVA; Mean Difference (Final Values) = -17.4, 95% CI 2-sided [-21.2 to -10.1]
Statistical Analysis 2: Comparison: Amlodipine vs Placebo; Test type: Superiority or Other; p = 0.001, ANOVA; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-17.4 to -6.3]

4. Primary Outcome: Change From Baseline (0 Hours) to Week 4 in Central SBP After Multiple Doses of Treatment
Description: Central SBP was measured by the SphygmoCor® device. Central SBP was measured at baseline and at 24 hours post dose on Day 28 (Week 4) and expressed as a change from baseline.
Time Frame: Baseline (0 hrs), 24 hours after the Day 28 dose
Population: 33 participants completed all study periods and provided more than 1 period of BP data, and were thus evaluable for the BP analyses.
  Unreliable SphygmoCor® data were collected for one participant in the ISM ER treatment group, therefore this participant was excluded from the multiple dose SBP analysis.
Measure: Least Squares Mean (Standard Deviation); unit: mm mercury (Hg)
Arm/Group | ISMN ER | Amlodipine | Placebo
Number analyzed (Participants) | 32 | 33 | 33
mm mercury (Hg) | -0.7 (11.6) | -12.9 (11.6) | 3.2 (11.6)
Statistical Analysis 1: Comparison: ISMN ER vs Placebo; Test type: Superiority or Other; p = 0.186, ANOVA; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-9.5 to 1.8]
Statistical Analysis 2: Comparison: Amlodipine vs Placebo; Test type: Superiority or Other; p < 0.0005, ANOVA; Mean Difference (Final Values) = -16.1, 95% CI 2-sided [-21.7 to -10.5]

5. Primary Outcome: TWA Change From Baseline (0 Hours) to 12 Hours in Central Diastolic Blood Pressure (DBP) After A Single Dose of Treatment
Description: Central DBP was measured by the SphygmoCor® device. Single dose effects on central DBP were estimated as a time-weighted average change from baseline over the 12-hour post single dose observation period.
Time Frame: Baseline (0 hrs), 12 hours post-dose (Day 1)
Population: 33 participants completed all study periods and provided more than 1 period of BP data, and were thus evaluable for the BP analyses.
  Unreliable SphygmoCor® data were collected for one participant in the ISM ER treatment group, therefore this participant was excluded from the single dose DBP analysis.
Measure: Least Squares Mean (Standard Deviation); unit: mm mercury (Hg)
Arm/Group | ISMN ER | Amlodipine | Placebo
Number analyzed (Participants) | 32 | 33 | 33
mm mercury (Hg) | -8.2 (5.9) | -2.1 (5.9) | 1.1 (5.9)
Statistical Analysis 1: Comparison: ISMN ER vs Placebo; Test type: Superiority or Other; p < 0.0005, ANOVA; Median Difference (Final Values) = -9.2, 95% CI 2-sided [-12.1 to -6.4]
Statistical Analysis 2: Comparison: Amlodipine vs Placebo; Test type: Superiority or Other; p = 0.035, ANOVA; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-6.0 to -0.3]

6. Primary Outcome: Change From Baseline (0 Hours) to Week 4 in Central DBP After Multiple Doses of Treatment
Description: Central DBP was measured by the SphygmoCor® device. Central DBP was measured at baseline and at 24 hours post dose on Day 28 (Week 4) and expressed as a change from baseline.
Time Frame: Baseline (0 hrs), 24 hours after the Day 28 dose
Population: 33 participants completed all study periods and provided more than 1 period of BP data, and were thus evaluable for the BP analyses.
  Unreliable SphygmoCor® data were collected for one participant in the ISM ER treatment group, therefore this participant was excluded from the multiple dose DBP analysis.
Measure: Least Squares Mean (Standard Deviation); unit: mm mercury (Hg)
Arm/Group | ISMN ER | Amlodipine | Placebo
Number analyzed (Participants) | 32 | 33 | 33
mm mercury (Hg) | -0.7 (9.0) | -7.7 (9.0) | 1.1 (9.0)
Statistical Analysis 1: Comparison: ISMN ER vs Placebo; Test type: Superiority or Other; p = 0.428, ANOVA; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-6.1 to 2.6]
Statistical Analysis 2: Comparison: Amlodipine vs Placebo; Test type: Superiority or Other; p < 0.0005, ANOVA; Mean Difference (Final Values) = -8.8, 95% CI 2-sided [-13.1 to -4.5]

7. Primary Outcome: TWA Change From Baseline (0 Hours) to 12 Hours in Peripheral SBP After A Single Dose of Treatment
Description: Peripheral SBP was measured by Brachial Sphygmomanometer (standard cuff). Single dose effects on peripheral SBP were estimated as a time-weighted average change from baseline over the 12-hour post single dose observation period.
Time Frame: Baseline (0 hrs), 12 hours post-dose (Day 1)
Population: 33 participants completed all study periods and provided more than 1 period of BP data, and were thus evaluable for the BP analyses.
Measure: Least Squares Mean (Standard Deviation); unit: mm mercury (Hg)
Arm/Group | ISMN ER | Amlodipine | Placebo
Number analyzed (Participants) | 33 | 33 | 33
mm mercury (Hg) | -12.1 (7.7) | -3.1 (7.7) | 1.7 (7.7)
Statistical Analysis 1: Comparison: ISMN ER vs Placebo; Test type: Superiority or Other; p < 0.0005, ANOVA; Mean Difference (Final Values) = -13.7, 95% CI 2-sided [-17.5 to -10.0]
Statistical Analysis 2: Comparison: Amlodipine vs Placebo; Test type: Superiority or Other; p = 0.015, ANOVA; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-8.5 to -1.0]

8. Primary Outcome: Change From Baseline (0 Hours) to Week 4 in Peripheral SBP After Multiple Doses of Treatment
Description: Peripheral SBP was measured by Brachial Sphygmomanometer (standard cuff). Peripheral SBP was measured at baseline and at 24 hours post dose on Day 28 (Week 4) and expressed as a change from baseline.
Time Frame: Baseline (0 hrs), 24 hours after the Day 28 dose
Population: as for outcome 7
Measure: Least Squares Mean (Standard Deviation); unit: mm mercury (Hg)
Arm/Group | ISMN ER | Amlodipine | Placebo
Number analyzed (Participants) | 33 | 33 | 33
mm mercury (Hg) | -0.6 (11.2) | -11.4 (11.2) | 3.9 (11.2)
Statistical Analysis 1: Comparison: ISMN ER vs Placebo; Test type: Superiority or Other; p = 0.112, ANOVA; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-9.9 to 1.0]
Statistical Analysis 2: Comparison: Amlodipine vs Placebo; Test type: Superiority or Other; p < 0.0005, ANOVA; Mean Difference (Final Values) = -15.3, 95% CI 2-sided [-20.7 to -9.8]

9. Primary Outcome: TWA Change From Baseline (0 Hours) to 12 Hours in Peripheral DBP After A Single Dose of Treatment
Description: Peripheral DBP was measured by Brachial Sphygmomanometer (standard cuff). Single dose effects on peripheral DBP were estimated as a time-weighted average change from baseline over the 12-hour post single dose observation period.
Time Frame: Baseline (0 hrs), 12 hours post-dose (Day 1)
Population: as for outcome 7
Measure: Least Squares Mean (Standard Deviation); unit: mm mercury (Hg)
Arm/Group | ISMN ER | Amlodipine | Placebo
Number analyzed (Participants) | 33 | 33 | 33
mm mercury (Hg) | -8.0 (5.7) | -2.0 (5.7) | 1.0 (5.7)
Statistical Analysis 1: Comparison: ISMN ER vs Placebo; Test type: Superiority or Other; p < 0.0005, ANOVA; Mean Difference (Final Values) = -9.0, 95% CI 2-sided [-11.8 to -6.2]
Statistical Analysis 2: Comparison: Amlodipine vs Placebo; Test type: Superiority or Other; p = 0.039, ANOVA; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-5.8 to -0.2]

10. Primary Outcome: Change From Baseline (0 Hours) to Week 4 in Peripheral DBP After Multiple Doses of Treatment
Description: Peripheral SBP was measured by Brachial Sphygmomanometer (standard cuff). Peripheral DBP was measured at baseline and at 24 hours post dose on Day 28 (Week 4) and expressed as a change from baseline.
Time Frame: Baseline (0 hrs), 24 hours after the Day 28 dose
Population: as for outcome 7
Measure: Least Squares Mean (Standard Deviation); unit: mm mercury (Hg)
Arm/Group | ISMN ER | Amlodipine | Placebo
Number analyzed (Participants) | 33 | 33 | 33
mm mercury (Hg) | -1.4 (8.7) | -7.5 (8.7) | 1.0 (8.7)
Statistical Analysis 1: Comparison: ISMN ER vs Placebo; Test type: Superiority or Other; p = 0.267, ANOVA; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-6.6 to 1.8]
Statistical Analysis 2: Comparison: Amlodipine vs Placebo; Test type: Superiority or Other; p < 0.0005, ANOVA; Mean Difference (Final Values) = -8.5, 95% CI 2-sided [-12.7 to -4.3]

ADVERSE EVENTS:
Description: Adverse event data were unavailable for 4 participants in the Placebo treatment group and for 1 participant in the Amlodipine treatment group due to discontinuations during Period 1.
Arm/Group | Placebo | ISMN ER | Amlodipine
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 7/34 | 18/38 | 9/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=34) | ISMN ER (N=38) | Amlodipine (N=37)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 16 (16) | 6 (6)
Tension Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines